CLINICAL TRIAL: NCT03121573
Title: Efficacy and Safety of Duloxetine Among Individuals With Depressive Disorder in a 12 Weeks Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: SF14216
Record Dates: First submitted 2017-04-13; First posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
Keywords: near infrared spectroscopy, NIRS, duloxetine
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Other): medication: duloxetine 30 to 60 mg tablets by mouth, QD to BID.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — duloxetine 30 to 60 mg tablets by mouth, QD to BID per day,

SUMMARY:
The aim of this study was to investigate the effects of duloxetine on improvement of brain cortical activity in patients suffering from major depressive disorder using near infrared spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* HAMD-17 more than 12 points
* Participants could understand this study and sign permit
* Participants could receive NIRS measurements
* Participants could comply with the protocol of the study

Exclusion Criteria:

* alcohol or substance abuse within 3 months of the study
* ever participate other clinical study related to duloxetine
* previous poor treatment effects of duloxetine
* concomitant use of MAOi within 14 days
* concomitant use of Linezolid
* with uncontrolled glaucoma

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Change in Depression severity | 0-2-4-8-12 weeks
  Hamilton Rating Scale for Depression

SECONDARY OUTCOMES:
Change in Brain cortical activity | 0-2-4-8-12 weeks
  Using Near Infrared Spectroscopy

IPD SHARING:
Plan to Share IPD: No
no plan